CLINICAL TRIAL: NCT03952988
Title: Effect of the Consumption of a Probiotic (B. Bifidum 900791)-Containing Ice-cream in Adult With Hypolactasia and Lactose Intolerance
Brief Title: Effect of B.Bifidum 900791 Intake in Adult With Hypolactasia and Lactose Intolerance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Martin Gotteland, Head, Lab. of Digestive physiology, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UChile-Bifidice-2
Record Dates: First submitted 2019-04-08; First posted 2019-05-16 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Intervention Model Description: At Day 1, hypolactasic subjects will perform a Hydrogen Breath Test (HBT) with a placebo ice-cream with 20g lactose (Negative Control). A second HBT will be carried at Day-8 with the same product + an exogenous lactase (Positive control). A 3° HBT will be carried out at Day 15 with the probiotic ice cream with 20g lactose to determine the acute effect of the probiotic. Posteriorly, the subjects will be randomly assigned in one of 2 groups to consume an ice-cream/d, with or without the probiotic, for 4 weeks. At Day-43, they will carry out a 4° HBT with ice cream with 20g lactose and without probiotic (Evaluation of the chronic effect). At Day 71, after 4 weeks washout period, a 5° HBT will be carried out with the ice cream with lactose and without probiotic, to evaluate the remanence of the effect. A fresh stool will be obtained at days 15, 43 and 71 to determine the presence of the probiotic, microbiota composition, ß-galactosidase activity and short chain fatty acid concentrations.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental)
  Interventions: Dietary Supplement: Probiotic ice cream
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo ice cream

INTERVENTIONS:
Dietary Supplement: Probiotic ice cream — One portion (50g) of an ice-cream containing the probiotic B. bifidum 900791 (>10(exp7)/g) every day for 4 weeks
  Other Names: Bifidice
  Arms: Probiotic
Dietary Supplement: Placebo ice cream — One portion (50g) of an ice-cream without probiotic every day for 4 weeks
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Lactase is high in the newborn intestine, allowing him to digest the high amounts of lactose present in breastmilk. From weaning, lactase is genetically programmed to decrease, reaching residual levels in the adult. This situation occurs in 75% of the world population and is known as "adult primary hypolactasia" while the remaining 25% is "lactase persistent" i.e. maintains in adulthood lactase values similar to these of newborns. In subjects with hypolactasia, the intake of milk products can produce digestive symptoms, making that the affected individuals spontaneously reduce the consumption of these products and, therefore, their intake of calcium and proteins.

In addition to lactose-free milk and exogenous lactase, a strategy for the intolerant subjects to continue consuming dairy products is, for example, to consume yogurt, due to the fact that the lactase of the yogurt bacteria continues to function in the intestine of the consumer, hydrolyzing lactose and decreasing the development of digestive symptoms. Similarly, many probiotic strains, such as L. acidophilus NCFM, L. casei CRL431, B. longum 401 and B. bifidum Orla Jensen 1424, express β-galactosidases that hydrolyze lactose, preventing its fermentation and the production of gases. The acute administration of these strains improves lactose tolerance. In addition, a recent study reported that dietary supplementation of intolerant subjects for 4 weeks with L. casei Shirota and B. breve Yakult reduced digestive symptoms and breath hydrogen excretion not only at the end of the period of administration of the probiotics but also 3 months after having discontinued the use of probiotics.

Based on this background, the aim of this study is to determine whether the regular consumption of an ice cream with the strain B. bifidum 900791 improves lactose intolerance in hypolactasic subjects, even after the suspension of the consumption of the product. To determine if this effect is due to the adaptation of the microbiota, the investigators will also evaluate changes in the composition of the microbiota and the generation of volatile fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypolactasia and lactose intolerance

Exclusion Criteria:

* Diarrhea
* Previous gastrointestinal pathologies
* Current or recent intake of antibiotics, anti-inflammatory drugs, laxatives or drugs interfering with intestinal transit
* Alterations of intestinal anatomy or function
* Pregnancy
* Chronic diseases of different etiologies (auto-immune, inflammatory, tumor, etc.).

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Area under curve (AUC) of hydrogen in the HBT | Day 15
  Acute effect of the probiotic on hydrogen excretion after lactose ingestion

SECONDARY OUTCOMES:
Area under curve (AUC) of hydrogen in the HBT | Day 43
  Chronic effect of the probiotic on hydrogen excretion after lactose ingestion
Area under curve (AUC) of hydrogen in the HBT | Day 71
  Remanent effect of the probiotic on hydrogen excretion after lactose ingestion after one month without probiotic ingestion
Fecal microbiota alpha-diversity | Days 15
  Shannon Index
Fecal microbiota alpha-diversity | Day 43
  Shannon Index
Fecal microbiota alpha-diversity | Day 71
  Shannon Index
Relative abundancies of the bacterial taxa forming the the fecal microbiota | Day 15
  Relative abundancies of the different bacterial taxa detected by high throughput sequencing
Relative abundancies of the bacterial taxa forming the the fecal microbiota | Day 43
  Relative abundancies of the different bacterial taxa detected by high throughput sequencing
Relative abundancies of the bacterial taxa forming the the fecal microbiota | Day 71
  Relative abundancies of the different bacterial taxa detected by high throughput sequencing
Fecal counts of B. bifidum 900791 | Days 15
  B. bifidum 900791 counts in fecal samples
Fecal counts of B. bifidum 900791 | Days 43
  B. bifidum 900791 counts in fecal samples
Fecal counts of B. bifidum 900791 | Days 71
  B. bifidum 900791 counts in fecal samples
Fecal beta-galactosidase activity | Days 15
  Determination of the microbial beta-galactosidase activity in fecal samples (expressed as U/g)
Fecal beta-galactosidase activity | Days 43
  Determination of the microbial beta-galactosidase activity in fecal samples (expressed as U/g)
Fecal beta-galactosidase activity | Days 71
  Determination of the microbial beta-galactosidase activity in fecal samples (expressed as U/g)
Fecal short chain fatty acids concentrations | Days 15
  Determination of short chain fatty acids concentrations in fecal samples
Fecal short chain fatty acids concentrations | Days 43
  Determination of short chain fatty acids concentrations in fecal samples
Fecal short chain fatty acids concentrations | Days 71
  Determination of short chain fatty acids concentrations in fecal samples
Scores of gastrointestinal symptoms: bloating, abdominal distention, abdominal pain, borborygms and flatulence, during the HBT | Days 15
  Determination of gastrointestinal symptoms (bloating, abdominal distention, abdominal pain, borborygms and flatulence) using a previously validated questionnaire on a scale of 0 (none), 1 (mild), 2 (moderate), 3 (severe). We will define clinically relevant ymptoms as a composite score of 3 or more during the HBT.
Scores of gastrointestinal symptoms: bloating, abdominal distention, abdominal pain, borborygms and flatulence, during the HBT | Days 43
  Determination of gastrointestinal symptoms (bloating, abdominal distention, abdominal pain, borborygms and flatulence) using a previously validated questionnaire on a scale of 0 (none), 1 (mild), 2 (moderate), 3 (severe). We will define clinically relevant ymptoms as a composite score of 3 or more during the HBT.
Scores of gastrointestinal symptoms: bloating, abdominal distention, abdominal pain, borborygms and flatulence, during the HBT | Days 71
  Determination of gastrointestinal symptoms (bloating, abdominal distention, abdominal pain, borborygms and flatulence) using a previously validated questionnaire on a scale of 0 (none), 1 (mild), 2 (moderate), 3 (severe). We will define clinically relevant ymptoms as a composite score of 3 or more during the HBT.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marteau P, Pochart P, Flourie B, Pellier P, Santos L, Desjeux JF, Rambaud JC. Effect of chronic ingestion of a fermented dairy product containing Lactobacillus acidophilus and Bifidobacterium bifidum on metabolic activities of the colonic flora in humans. Am J Clin Nutr. 1990 Oct;52(4):685-8. doi: 10.1093/ajcn/52.4.685. PMID 2119557
- [Result] Pelletier X, Laure-Boussuge S, Donazzolo Y. Hydrogen excretion upon ingestion of dairy products in lactose-intolerant male subjects: importance of the live flora. Eur J Clin Nutr. 2001 Jun;55(6):509-12. doi: 10.1038/sj.ejcn.1601169. PMID 11423928
- [Result] Jiang T, Mustapha A, Savaiano DA. Improvement of lactose digestion in humans by ingestion of unfermented milk containing Bifidobacterium longum. J Dairy Sci. 1996 May;79(5):750-7. doi: 10.3168/jds.S0022-0302(96)76422-6. PMID 8792277
- [Result] Almeida CC, Lorena SL, Pavan CR, Akasaka HM, Mesquita MA. Beneficial effects of long-term consumption of a probiotic combination of Lactobacillus casei Shirota and Bifidobacterium breve Yakult may persist after suspension of therapy in lactose-intolerant patients. Nutr Clin Pract. 2012 Apr;27(2):247-51. doi: 10.1177/0884533612440289. Epub 2012 Mar 8. PMID 22402407
- [Result] Turroni F, Duranti S, Bottacini F, Guglielmetti S, Van Sinderen D, Ventura M. Bifidobacterium bifidum as an example of a specialized human gut commensal. Front Microbiol. 2014 Aug 21;5:437. doi: 10.3389/fmicb.2014.00437. eCollection 2014. PMID 25191315
- [Result] Gargari G, Taverniti V, Balzaretti S, Ferrario C, Gardana C, Simonetti P, Guglielmetti S. Consumption of a Bifidobacterium bifidum Strain for 4 Weeks Modulates Dominant Intestinal Bacterial Taxa and Fecal Butyrate in Healthy Adults. Appl Environ Microbiol. 2016 Sep 16;82(19):5850-9. doi: 10.1128/AEM.01753-16. Print 2016 Oct 1. PMID 27451450
- [Result] Hsu CA, Yu RC, Lee SL, Chou CC. Cultural condition affecting the growth and production of beta-galactosidase by Bifidobacterium longum CCRC 15708 in a jar fermenter. Int J Food Microbiol. 2007 May 1;116(1):186-9. doi: 10.1016/j.ijfoodmicro.2006.12.034. Epub 2007 Jan 19. PMID 17320993